CLINICAL TRIAL: NCT00559559
Title: PAtient NOtifier Feature for Reduction of Anxiety: A Multicenter ICD Study
Brief Title: PAtient NOtifier Feature for Reduction of Anxiety
Acronym: Panoramic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CR06002HV
Record Dates: First submitted 2007-11-15; First posted 2007-11-16 (Estimated); Last update posted 2019-02-04 (Actual); Status verified 2019-02

CONDITIONS: Tachycardia, Ventricular
Keywords: Primary and secondary prevention for ventricular tachycardia
MeSH Terms: conditions — Tachycardia, Ventricular | interventions — Defibrillators, Implantable

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Group (Other): Patient Notifier turned OFF
  Interventions: Device: ICD implant + Patient Notifier turned OFF
- Treatment group (Experimental): Patient Notifier turned ON
  Interventions: Procedure: ICD Implant + Patient Notifier turned ON

INTERVENTIONS:
Device: ICD implant + Patient Notifier turned OFF — ICD implant, plus standard care, i.e. Patient Notifier turned off
  Arms: Control Group
Procedure: ICD Implant + Patient Notifier turned ON — ICD implant. The Patient Notifier™ feature will be turned ON.
  Arms: Treatment group

SUMMARY:
This study is intended to look at the effect of the SJM vibrating Patient Notifier™ system, which will warn the patient of possible failures of the implanted system, on reducing patient device related anxiety

ELIGIBILITY:
Inclusion Criteria:

* Patient has recently (min. 2 weeks - max. 14 weeks) been implanted with an SJM ICD with the Patient Notifier™ feature;
* Patient is willing and able to independently comprehend and complete the study-related questionnaires;
* Patient has signed the study specific informed consent form.

Exclusion Criteria:

* have already had a Patient Notifier™ alert since implant;
* had a prior device implant (PM or ICD);
* have not been discharged from the hospital since device implant;
* have evidence of psychosis, dementia or cognitive impairment as documented in the patients' hospital records;
* cannot commit to the follow-up schedule;
* have a life expectancy of less than 1 year;
* are on a waiting list for a heart transplant;
* are less than 18 years old;
* are pregnant;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 362 (Actual)
Dates: Start 2007-12; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Reduction in device related anxiety, related to battery depletion, as assessed by the Duru Questionnaire (question 9) Reduction in device related anxiety, related to device malfunction, as assessed by the Duru Questionnaire (question 10) | 12months

SECONDARY OUTCOMES:
Reduction in general anxiety Evolution over time in anxiety for the different personality types Cross-overs Sensitivity and Specificity of the Patient Notifier™ Number of appropriate/inappropriate ICD therapies Hospitalizations Mortality | 1year

CONTACTS AND LOCATIONS:
Overall Officials: Firat Duru, Prof., Principal Investigator — Universitätsspital Zürich
Locations (1):
- UniversitätsSpital Zürich, Zurich, Switzerland

REFERENCES:
- [Derived] Duru F, Dorian P, Favale S, Perings C, Pedersen SS, Willems V; PAtient NOtifier Feature for Reduction of Anxiety: A Multicenter ICD Study investigators. Effects of an alert system on implantable cardioverter defibrillator-related anxiety: rationale, design, and endpoints of the PANORAMIC multicentre trial. Europace. 2010 May;12(5):726-30. doi: 10.1093/europace/euq026. Epub 2010 Mar 5. PMID 20207746